CLINICAL TRIAL: NCT02386202
Title: Augmented Renal Clearance in Hemorrhagic Stroke Patients Admitted to the Neurosciences Intensive Care Unit
Brief Title: ARC in Hemorrhagic Stroke
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1491
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Hemorrhagic Stroke; Augmented Renal Clearance
MeSH Terms: conditions — Hemorrhagic Stroke

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with hemorrhagic stroke: All patients with hemorrhagic stroke admitted to the neurosciences ICU are eligible for study enrollment.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No interventions

SUMMARY:
To determine the incidence and predictors of augmented renal clearance (ARC) in patients with hemorrhagic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* Patients with hemorrhagic stroke
* Anticipated length of stay in the neuroscience intensive care unit > 48 hours
* Informed consent provided by the patient or by the patient's designated medical proxy

Exclusion Criteria:

* Pregnancy
* Patients with pre-existing renal dysfunction (chronic kidney disease stages 3 - 5)
* Patients receiving renal replacement therapy
* Patients with an admission serum creatinine > 1.4 mg/dL
* Patients with non-aneurysmal subarachnoid hemorrhage
* Patients with history of nephrectomy or body mass index < 18 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients with hemorrhagic stroke admitted to the University of North Carolina Neurosciences Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To describe the onset, magnitude, and change over time of ARC in patients with hemorrhagic stroke | Over neurosciences intensive care unit stay
  Daily 8-hour urine collections will be performed to directly measure creatinine clearance up to ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A Morbitzer, PharmD, Principal Investigator — UNC Eshelman School of Pharmacy
Locations (1):
- University of North Carolina Hospitals, Chapel Hill, North Carolina, United States